CLINICAL TRIAL: NCT01153022
Title: Effect of Joint Mobilization on Alpha Motoneuron Reflex Excitability in People With Spasticity: Controlled Clinical Trial
Brief Title: Effect of Joint Mobilization on Alpha Motoneuron Reflex Excitability
Acronym: JM-HRreflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Manizales, Colombia (Other)
Responsible Party: María del Carmen Vergara Quintero, Universidad Autónoma de Manizales
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CT01UAM-H reflex
Record Dates: First submitted 2010-05-12; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Muscle Spasticity; Spinal Cord Injury; Stroke; Craniocerebral Trauma
Keywords: Musculoskeletal manipulations; Muscle spasticity
MeSH Terms: conditions — Muscle Spasticity; Spinal Cord Injuries; Stroke; Craniocerebral Trauma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: joint mobilization techniques — In the experimental group, ankle joint mobilization was applied for five minutes, using grade II joint traction rhythmic oscillation (Mailland Scale) with the knee in 15° of flexion, subtalar in neutral and ankle in resting position (10º plantarflexion). During the control study, participants were placed under the same conditions as those of the experimental group but only the hands of the evaluator were placed in the foot, in the position of joint traction simulation.

SUMMARY:
Objective: To determine the effect of ankle joint mobilization on the alpha motoneuron reflex excitability of the soleus muscle in people with spasticity.

Subjects and Methods: A controlled clinical trial with crossover design and simple masking was conducted in 24 randomized subjects to initiate the control or experimental group. Traction and rhythmic oscillation were applied for five minutes to the ankle joint. Alpha motoneuron reflex excitability was assessed by measuring H wave amplitude (Hoffmann reflex - H reflex), stimulating the tibial nerve at the level of the popliteal fossa and recording in the soleus muscle. In each subject 12 measurements were taken: basal rate, during and after mobilization. Changes in alpha motoneuron reflex excitability were calculated in relation to basal measurement. For each measurement a hypothesis test was performed (Student t test).

Results: In groups of patients with brain injury (BI) and incomplete spinal cord injury (ISCI), a significant difference was found between measurements of both studies, concerning variation in alpha motoneuron reflex excitability during the application of joint mobilization techniques, with a decrease in the experimental group and an increase in the control group. In contrast, no significant differences were found after mobilization therapy. Patients with complete spinal cord injury (CSCI) showed no significant differences in any measurements.

Conclusion: We demonstrate the effectiveness of passive movement in the decrease of muscle tone during the mobilization maneuver in patients with BI or ISCI, but no residual effect after completion of the trial. This research project showed no evidence regarding spasticity reduction in complete spinal cord injuries. This suggests that therapeutic interventions to decrease muscle tone, based on the passive exercise and stimulation of proprioceptors should be reconsidered.

ELIGIBILITY:
Inclusion criteria:

* people over 18 years old
* spasticity acquired after five years of age
* any etiology
* any location of the injury

Patients were instructed not to consume coffee, cigarettes or energy drinks 24 hours prior to the study nor participate in excessive physical exercise during the day.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
H reflex | Twelve measurements were performed for each patient: basal rate (0), during joint mobilization (1, 3 and 5 minutes) and after the completion of joint mobilization (1, 3, 5, 10, 15, 20, 25 and 30 minutes)
  The Hoffmann reflex is an electrically induced reflex, analogous to the myotatic reflex that is mechanically triggered by stretching the neuromuscular spindle. In contrast, the H reflex stimulates the Ia fiber at the peripheral nerve level.

CONTACTS AND LOCATIONS:
Overall Officials: Julio E Pérez, Master, Principal Investigator — Universidad Autónoma de Manizales
Locations (1):
- UAM, Manizales, Caldas Department, Colombia